CLINICAL TRIAL: NCT00882011
Title: Observational Controlled Clinical Trials, on Adult Patients With T-lymphoblastic Lymphoma Treated With Intensive Chemo/Radiotherapy or Intensive Chemotherapy Followed by Transplant. Evaluation of Clinical, Anatomy-pathological Parameters
Brief Title: Observational Controlled Clinical Trials, on Adult Patients With T-lymphoblastic Lymphoma Treated With Intensive Chemo/Radiotherapy or Intensive Chemotherapy Followed by Transplant. Evaluation of Clinical, Anatomy -Pathological Parameters
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Fondazione Italiana Linfomi - ETS (Other)
Responsible Party: Sponsor
Other Study IDs: IIL-LY_01
Record Dates: First submitted 2009-04-15; First posted 2009-04-16 (Estimated); Last update posted 2011-10-13 (Estimated); Status verified 2011-10

CONDITIONS: Lymphoblastic Lymphoma
Keywords: T-lymphoblastic lymphoma; Intensive chemo/radiotherapy; Intensive chemotherapy; Transplant; Adult patients
MeSH Terms: conditions — Precursor Cell Lymphoblastic Leukemia-Lymphoma; Precursor T-Cell Lymphoblastic Leukemia-Lymphoma | interventions — Transplantation

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — Involved lymph nodes biopsy; biopsies performed in other areas affected by lymphoma; bone marrow blood; peripheral blood.
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- Arm 1: Adult patients with T-lymphoblastic lymphoma treated with intensive chemo/radiotherapy or intensive chemotherapy followed by transplant.
  Interventions: Other: Latest generation chemotherapies for T-LBL + transplant

INTERVENTIONS:
Other: Latest generation chemotherapies for T-LBL + transplant — 1. Standard doses of one of the following chemotherapies:
     * Holzer
     * LSA2-L2 modified
     * Stanford regimen
     * Hyper CVAD
     * Sequential treatments analogous to the ones above mentioned (e.g.: GIMEMA LAL094, others)
     * Intensive chemotherapy, ALL-type, MRD oriented (NILG-TLL Clinical Trial)
  2. Autologous transplant or allogeneic transplant or mini-allogeneic transplant

SUMMARY:
The purpose of the study is to create a prospective database of T-Lymphoblastic Lymphoma (T-LBL) cases in order to conduct an appropriate statistical study as well as to monitor diagnosis and minimal residual disease (MRD), to detect specific genetic profile useful to give advices on therapies, to assess if PET has a prognostic validity on T-Lymphoblastic Lymphoma (T-LBL).

DETAILED DESCRIPTION:
Observational prospective Clinical Trial designed to:

* record all patients treated with a latest generation ALL-like therapy (e.g.: Holzer, LSA2-L2 modified, GIMEMA LAL094), an enhanced therapy (hyper-CVAD or Stanford), autologous or allogeneic transplant or reduced intensity conditioning allotransplant after induction/consolidation and also expected cases treated with high dose sequential therapy or intensified minimal residual disease (MRD) oriented therapy;
* enter classic T-LBL patients (bone marrow infiltrate <25%) treated as long as previous section;
* monitor therapy response/phenotype ratio by the study of phenotype;
* monitor therapy response/residual disease/patients outcome ratio by the study of T-cell receptor gene rearrangement;
* evaluate any gene-profile difference between T-LBL pre-thymic phenotype and T-LBL thymic phenotype so as to correlate it to outcome;
* monitor the stage of the disease at diagnosis, during the therapy and during the follow-up by means of TAC, so to value if PET (in association with TAC) is an additional and/or outcome predicting element compared to TAC.

ELIGIBILITY:
Inclusion Criteria:

* no previous therapy, except for treatments to face up to clinical presentation of emergency;
* medical history initially characterized by nodal mass/masses;
* histological and immunophenotypic diagnosis that documents the diagnosis of T-LBL; in cases of bone marrow involvement and difficulties in obtaining nodal material, diagnosis could be based on bone marrow;
* availability of biological material for the study of TCR and gene-profile;
* age ≥ 15 years;
* all stages;
* infiltrated bone marrow <25%;
* normal liver, renal and cardiac functions, except for alterations directly related to lymphoma;
* estimates of treatment according to one of the last generation schedules;
* written informed consent.

Exclusion Criteria:

* patients with previous HCV, HBsAg+ or suffering from HIV;
* patients with organic pathology not related to lymphoma.

Min Age: 15 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: Adult patients with T-lymphoblastic lymphoma treated with intensive chemo/radiotherapy or intensive chemotherapy followed by transplant.
Sampling Method: Probability Sample
Enrollment: 100 (Estimated)
Dates: Start 2009-04; Primary Completion 2014-04 (Estimated); Study Completion 2019-04 (Estimated)

PRIMARY OUTCOMES:
To create a prospective database of T-lymphoblastic lymphoma cases on adult patients in order to conduct an appropriate statistical study. | 5 years

SECONDARY OUTCOMES:
To monitor histological and immunophenotypical diagnosis and to make a minimal residual disease (MRD) molecular study in order to verify if minimal residual disease (MRD) prognostic value observed in children is confirmed in adult patients. | 5 years
To make a gene expression analysis on T-Lymphoblastic Lymphoma patients to detect specific genetic profiles useful to give prognostic and therapy response advices. | 5 years
To validated the prognostic systems already identified in T-Acute Lymphoblastic Leukemia cases that can be useful to label the high-risk for Lymphoblastic Lymphoma patients. | 5 years
To evaluate if PET has a prognostic value in T-Lymphoblastic Lymphoma cases. | 5 years

CONTACTS AND LOCATIONS:
Overall Officials: Massimo Federico, MD, Study Director — Azienda Ospedaliero-Universitaria di Modena (MO)
Locations (16):
- Italy (16):
  - Ospedale dell'Angelo, Mestre, VE
  - Casa Sollievo della Sofferenza, Foggia
  - Ospedale San Martino, Genova
  - Ospedale Vito Fazzi, Lecce
  - Azienda Ospedaliera Papardo, Messina
  - Università degli studi di Modena, Modena
  - Policlinico San Matteo, Pavia
  - Ospedale Civile Santo Spirito, Pescara
  - Ospedale San Carlo, Potenza
  - Ospedale Bianche Melacrino Morelli, Reggio Calabria
  - Ospedale Sant'Eugenio, Roma
  - Università La Sapienza, Roma
  - Azienda Ospedaliera Sassari, Sassari
  - Ospedale San Giovanni Battista Molinette, Torino
  - San Giovanni Battista Molinette - Biologia Molecolare, Torino
  - Policlinico GB Rossi, Verona